CLINICAL TRIAL: NCT03102242
Title: Phase II Trial of Induction Immunotherapy With Atezolizumab for Patients With Unresectable Stage IIIA and IIIB NSCLC Eligible for Chemoradiotherapy With Curative Intent.
Brief Title: Atezolizumab Immunotherapy in Patients With Advanced NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFT-16
Record Dates: First submitted 2017-03-27; First posted 2017-04-05 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Induction immunotherapy: atezolizumab 1200 mg IV q 21 days x 4 cycles. Restaging after cycle 2 and cycle 4 induction: patients with progression of disease (PD) at the post-cycle 2 assessment will stop atezolizumab and go immediately to chemoradiotherapy if still stage III and eligible for curative intent therapy.
  Chemoradiotherapy: carboplatin AUC = 2 + paclitaxel 50 mg/m2 IV weekly x 6 weeks concurrent with radiation to a total dose of 60 Gy given in 2 Gy fractions daily M-F x 30 fractions
  Consolidation chemotherapy: Carboplatin AUC = 6 + paclitaxel 200 mg/m2 IV q 21 days x 2 cycles beginning 3-5 weeks after completion of radiation.
  Adjuvant immunotherapy: atezolizumab 1200 mg IV q 21 days to complete one year of therapy (from start of induction).
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Single arm phase II trial of induction immunotherapy with anti-PD-L1 for patients with unresectable stage III NSCLC and PS 0-1.

SUMMARY:
Phase II trial of induction immunotherapy with atezolizumab for patients with unresectable stage IIIA and IIIB NSCLC eligible for chemoradiotherapy with curative intent.

DETAILED DESCRIPTION:
This phase II pilot trial will combine neoadjuvant immunotherapy with Atezolizumab q 21 days for 12 weeks with standard chemoradiotherapy with curative intent for good PS patients with unresectable stage IIIA/B NSCLC. Because of the consequences of progression in this curative-intent population, restaging CT scans will be carried out after the first 2 cycles of neoadjuvant therapy. Non progressing patients will complete a total of one year of anti-PDL1 therapy with an interruption during chemoradiotherapy. Patients with evidence of progression at the first restaging evaluation will proceed immediately to chemoradiotherapy if still eligible for curative intent therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage IIIA/B NSCLC, PS 0-1
* No active autoimmune disease or uncontrolled infection, normal bone marrow, renal, hepatic function, FEV1 > 1.2L, no significant underlying heart or lung disease
* Pathologically proven diagnosis of NSCLC
* Measurable Stage IIIA or IIIB disease
* Tissue available for PD-L1 testing and for correlative science testing
* Patients must be considered unresectable or inoperable. Patients with nodal recurrence after surgery for early-stage NSCLC are eligible if the following criteria are met:

  * No prior chemotherapy or radiation for this lung cancer.
  * Prior curative-intent surgery at least 3 months prior to the nodal recurrence.
* Stage III A or B disease with minimum diagnostic evaluation within 6 weeks to include:

  * History/physical examination
  * Contrast enhanced CT of the chest and upper abdomen
  * MRI of the brain with contrast (or CT with contrast if MRI is medically contraindicated)
  * PET/CT
* If pleural fluid is visible on CT scan thoracentesis to exclude malignancy should be obtained. Patients with effusions that are too small to tap are eligible.
* Patients must be at least 4 weeks from major surgery and must be fully recovered
* Age greater than or equal to 18 years.
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks or at least 4 unstained slides, with an associated pathology report, for central testing of tumor PD-L1 expression.

  * If an archived tumor block exists, then either the block or at least 4 unstained slides from the block should be submitted. Tumor tissue should be of good quality based on total and viable tumor content, i.e. at least 50 viable tumor cells and intact tissue architecture. Fine needle aspiration, brushing,and lavage samples are not acceptable. If the block is tissue from a core-needle biopsy, then the block should contain tissue from at least three cores to be sufficient for evaluation.
  * Patients who do not have existing (archived) tissue specimens meeting eligibility requirements may undergo a biopsy during the screening period. Acceptable samples include core needle biopsies for deep tumor tissue (minimum of three cores) or excisional, or forceps biopsies for endobronchial or nodal lesions. The tissue should be fixed in formalin and embedded on site and sent as a block.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1):

  * ANC ≥ 1500 cells/µL
  * WBC counts > 2500/µL
  * Lymphocyte count ≥ 300/µL
  * Platelet count ≥ 100,000/µL
  * Hemoglobin ≥ 10.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) with the following exception:
* Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.

  * AST and ALT ≤ 3.0 x ULN
  * Alkaline phosphatase ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation:
* (140 - age) x (weight in kg) x (0.85 if female)/ 72 x (serum creatinine in mg/dL)
* Measurable disease per RECIST v1.1 (see Appendix 3)
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use for 90 days after the last dose of Atezolizumab.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* INR and aPTT ≤ 1.5 x ULN • This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.

Exclusion Criteria:

* Active autoimmune disease
* Greater than minimal, exudative, or cytologically positive pleural effusions
* Involved contralateral hilar nodes
* 10% weight loss within the past month
* Known EGFR exon 19 or 21 mutation or ALK rearrangement
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; non-invasive conditions such as carcinoma in situ of the breast, localized prostate cancer, carcinoma in situ of the oral cavity, or cervix are all permissible.
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Prior severe infusion reaction to a monoclonal antibody
* Severe, active co-morbidity, defined as follows:
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, myocardial infarction within the last 6 months, uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration or within 2 weeks of cycle 1 day 1.
* Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, HIV testing is required for entry into this protocol due to the immunologic basis for induction treatment.
* Pregnancy, lactation, or inability or unwillingness to use medically acceptable forms of contraception if pregnancy is a risk.
* Any history of allergic reaction to paclitaxel or other taxanes, or to carboplatin;
* Uncontrolled neuropathy grade 2 or greater regardless of cause.
* Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment; however, the following are allowed:

  i. Hormone-replacement therapy or oral contraceptives ii. Herbal therapy > 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1)
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible.
* Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Inability to comply with study and follow-up procedures
* History of active autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis
* Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
* Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:
* Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
* Rash must cover less than 10% of body surface area (BSA)
* Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alcometasone dipropionate 0.05%)
* No acute exacerbations of underlying condition within the last 6 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Active tuberculosis
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study
* Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* Malignancies other than the disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate-specific antigen [PSA] ≤ 10 mg/mL, etc.)

Medication-Related Exclusion Criteria:

* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Ross, MD, Study Chair — Mayo Clinic; Monica Bertagnolli, MD, Principal Investigator — Alliance Foundation Trials
Locations (13):
- United States (13):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - UCSD Moores Cancer Center, La Jolla, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - EMMC Cancer Care, Brewer, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Metro MN Community Oncology Research Consortium, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Ohio State University James Cancer Center, Columbus, Ohio
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rizvi NA, Mazieres J, Planchard D, Stinchcombe TE, Dy GK, Antonia SJ, Horn L, Lena H, Minenza E, Mennecier B, Otterson GA, Campos LT, Gandara DR, Levy BP, Nair SG, Zalcman G, Wolf J, Souquet PJ, Baldini E, Cappuzzo F, Chouaid C, Dowlati A, Sanborn R, Lopez-Chavez A, Grohe C, Huber RM, Harbison CT, Baudelet C, Lestini BJ, Ramalingam SS. Activity and safety of nivolumab, an anti-PD-1 immune checkpoint inhibitor, for patients with advanced, refractory squamous non-small-cell lung cancer (CheckMate 063): a phase 2, single-arm trial. Lancet Oncol. 2015 Mar;16(3):257-65. doi: 10.1016/S1470-2045(15)70054-9. Epub 2015 Feb 20. PMID 25704439
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Reck M, Paz-Ares L. Immunologic checkpoint blockade in lung cancer. Semin Oncol. 2015 Jun;42(3):402-17. doi: 10.1053/j.seminoncol.2015.02.013. Epub 2015 Feb 19. PMID 25965358
- [Background] Tecentriq Package Insert, 06May 2016 http://www.accessdata.fda.gov/drugsatfda_docs/label/2016/761034s000lbl.pdf
- [Background] Johnson DB, Balko JM, Compton ML, Chalkias S, Gorham J, Xu Y, Hicks M, Puzanov I, Alexander MR, Bloomer TL, Becker JR, Slosky DA, Phillips EJ, Pilkinton MA, Craig-Owens L, Kola N, Plautz G, Reshef DS, Deutsch JS, Deering RP, Olenchock BA, Lichtman AH, Roden DM, Seidman CE, Koralnik IJ, Seidman JG, Hoffman RD, Taube JM, Diaz LA Jr, Anders RA, Sosman JA, Moslehi JJ. Fulminant Myocarditis with Combination Immune Checkpoint Blockade. N Engl J Med. 2016 Nov 3;375(18):1749-1755. doi: 10.1056/NEJMoa1609214. PMID 27806233
- [Background] Nishino M, Giobbie-Hurder A, Gargano M, Suda M, Ramaiya NH, Hodi FS. Developing a common language for tumor response to immunotherapy: immune-related response criteria using unidimensional measurements. Clin Cancer Res. 2013 Jul 15;19(14):3936-43. doi: 10.1158/1078-0432.CCR-13-0895. Epub 2013 Jun 6. PMID 23743568
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Derived] Ross HJ, Kozono D, Wang XF, Urbanic JJ, Williams TM, Nelson GD, Carbone DP, Chung D, Robb R, Byun WY, Talabere T, DuFrane C, Bara I, Schulze K, Brockman M, Gao J, Vokes EE, Stinchcombe TE. Atezolizumab Before and After Chemoradiation for Unresectable Stage III Non-Small Cell Lung Cancer: A Phase II Nonrandomized Controlled Trial. JAMA Oncol. 2024 Sep 1;10(9):1212-1219. doi: 10.1001/jamaoncol.2024.1897. PMID 39052256

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Treatment): Induction immunotherapy: atezolizumab 1200 mg IV q 21 days x 4 cycles. Restaging after cycle 2 and cycle 4 induction: patients with progression of disease (PD) at the post-cycle 2 assessment will stop atezolizumab and go immediately to chemoradiotherapy if still stage III and eligible for curative intent therapy.
Period: Overall Study
Arm/Group | Arm A (Treatment)
Started | 64
Completed | 62
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Arm A (Treatment)
Number analyzed (Participants) | 62
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.9 [57.7 to 71.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) After 12 Weeks Induction
Description: The primary objective of this single arm phase II trial is to determine whether neoadjuvant and adjuvant anti-PD-L1 therapy bracketing standard chemoradiation therapy and consolidation therapy is worthy of further investigation. The primary endpoint will be the disease control rate (DCR) after 12 weeks induction immunotherapy.
Time Frame: 12 weeks
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Treatment)
Number analyzed (Participants) | 62
proportion of participants | 0.742 [0.657 to 0.814]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is the rate of best overall response (complete or partial response) after 12 weeks of neoadjuvant atezolizumab therapy. ORR and its 90% Clopper-Pearson Confidence interval will be estimated.
Time Frame: 12 weeks
Population: Induction immunotherapy: atezolizumab 1200 mg IV q 21 days x 4 cycles. Restaging after cycle 2 and cycle 4 induction: patients with progression of disease (PD) at the post-cycle 2 assessment will stop atezolizumab and go immediately to chemoradiotherapy if still stage III and eligible for curative intent therapy.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Treatment)
Number analyzed (Participants) | 62
proportion of participants | 0.661 [0.573 to 0.761]

3. Secondary Outcome: Median PFS
Description: Progression-free survival (PFS) is defined as the time from the start of neoadjuvant therapy to disease progression or recurrence (first disease recurrence or death, whichever comes first). The Kaplan-Meier estimator will be used to estimate median PFS and confidence intervals.
Time Frame: 38.3 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Treatment)
Number analyzed (Participants) | 64
Months | 26.1 [15.8 to NA] — Not enough events to calculate upper interval.

4. Secondary Outcome: Progression Free Survival (PFS) at 12 and 24 Months
Description: Progression-free survival (PFS) is defined as the time from the start of neoadjuvant therapy to disease progression or recurrence (first disease recurrence or death, whichever comes first). The Kaplan-Meier estimator will be used to estimate median PFS and confidence intervals. A progression occurs when at least one of the following are true:
  1. At least one new malignant lesion, which also includes any lymph node that was normal at baseline (< 1.0 cm short axis) and increased to ≥ 1.0 cm short axis during follow-up.
  2. At least a 20% increase in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the MSD (Section 11.4.1). In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD.
  3. See Section 11.3.2 for details in regards to the requirements for PD via FDG-PET imaging.
Time Frame: 12 and 24 Months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Treatment)
Number analyzed (Participants) | 64
proportion of participants
  12 | 0.66 [0.56 to 0.79]
  24 | 0.5 [0.39 to 0.66]

5. Secondary Outcome: Median OS
Description: Overall Survival (OS) is defined as the time from the start of neoadjuvant therapy to death. The Kaplan-Meier estimator will be used to estimate median OS.
Time Frame: 38.3 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Treatment)
Number analyzed (Participants) | 64
Months | NA [NA to NA] — Not enough events for calculation of median or confidence intervals

6. Secondary Outcome: Overall Survival at 12 and 24 Months
Description: Overall Survival (OS) is defined as the time from the start of neoadjuvant therapy to death. The Kaplan-Meier estimator will be used to estimate OS at 12 months and 24 months, and their confidence intervals.
Time Frame: 12 and 24 Months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Treatment)
Number analyzed (Participants) | 64
proportion of participants
  12 months | 0.87 [0.79 to 0.96]
  24 months | 0.73 [0.62 to 0.85]

ADVERSE EVENTS:
Time Frame: 38.3 Months
Arm/Group | Arm A (Treatment)
All-Cause Mortality (participants affected / at risk) | 18/64
Serious Adverse Events (participants affected / at risk) | 34/64
Other Adverse Events (participants affected / at risk) | 59/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Treatment) (N=64)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Esophageal stenosis (Gastrointestinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 8 (8)
Sepsis (Infections and infestations) | 4 (5)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (5)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Treatment) (N=64)
Anemia (Blood and lymphatic system disorders) | 28 (74)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 6 (6)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 15 (15)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 5 (6)
Hypothyroidism (Endocrine disorders) | 7 (8)
Blurred vision (Eye disorders) | 8 (9)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 3 (3)
Floaters (Eye disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (19)
Bloating (Gastrointestinal disorders) | 5 (5)
Colitis (Gastrointestinal disorders) | 3 (6)
Constipation (Gastrointestinal disorders) | 26 (42)
Diarrhea (Gastrointestinal disorders) | 24 (46)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 15 (19)
Esophageal pain (Gastrointestinal disorders) | 2 (3)
Esophageal stenosis (Gastrointestinal disorders) | 2 (4)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 23 (31)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 11 (13)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 7 (14)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 (5)
Mucositis oral (Gastrointestinal disorders) | 8 (15)
Nausea (Gastrointestinal disorders) | 34 (46)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (4)
Stomach pain (Gastrointestinal disorders) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (24)
Chills (General disorders) | 11 (12)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 11 (18)
Edema trunk (General disorders) | 2 (4)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 42 (90)
Fever (General disorders) | 11 (12)
Flu like symptoms (General disorders) | 2 (3)
Gen disord and admin site conds-Oth spec (General disorders) | 3 (5)
Infusion site extravasation (General disorders) | 1 (1)
Localized edema (General disorders) | 2 (3)
Malaise (General disorders) | 1 (1)
Neck edema (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 16 (22)
Pain (General disorders) | 19 (31)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3)
Eye infection (Infections and infestations) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 6 (8)
Lung infection (Infections and infestations) | 7 (9)
Mucosal infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 10 (15)
Urinary tract infection (Infections and infestations) | 3 (4)
Vaginal infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Dermatitis radiation (Injury, poisoning and procedural complications) | 9 (11)
Fall (Injury, poisoning and procedural complications) | 4 (5)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (6)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (12)
Alkaline phosphatase increased (Investigations) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 14 (16)
Blood bilirubin increased (Investigations) | 3 (4)
Cardiac troponin I increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 7 (15)
ECG QT corrected interval prolonged (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
INR increased (Investigations) | 3 (3)
Investigations - Other, specify (Investigations) | 5 (5)
Lymphocyte count decreased (Investigations) | 19 (94)
Neutrophil count decreased (Investigations) | 8 (18)
Platelet count decreased (Investigations) | 15 (45)
Weight gain (Investigations) | 6 (13)
Weight loss (Investigations) | 12 (21)
White blood cell decreased (Investigations) | 18 (52)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 20 (30)
Dehydration (Metabolism and nutrition disorders) | 12 (13)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 11 (18)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (16)
Hyponatremia (Metabolism and nutrition disorders) | 13 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 (12)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 7 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (16)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 12 (14)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 7 (8)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 17 (22)
Lethargy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2)
Movements involuntary (Nervous system disorders) | 1 (2)
Muscle weakness right-sided (Nervous system disorders) | 1 (2)
Nervous system disorders - Oth spec (Nervous system disorders) | 4 (7)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 26 (37)
Presyncope (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 2 (3)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (4)
Agitation (Psychiatric disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 10 (10)
Depression (Psychiatric disorders) | 8 (9)
Insomnia (Psychiatric disorders) | 17 (20)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 3 (3)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (53)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 33 (66)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 (20)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 13 (35)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 12 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (29)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (10)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (22)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 6 (9)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 21 (39)
Hypotension (Vascular disorders) | 9 (12)
Phlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (5)
Vascular disorders - Other, specify (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03102242/Prot_SAP_000.pdf